CLINICAL TRIAL: NCT07180329
Title: Determination of Zinc and Selenium Bioactivity in Modulating Immune Parameters in Tuberculosis
Brief Title: Zinc and Selenium Bioactivity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lahore (Other)
Responsible Party: Principal Investigator, Sana Noreen, Assistant Professor, University of Lahore
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Supportive Care
Other Study IDs: REC-UOL-FAHS/906/2022
Record Dates: First submitted 2025-08-29; First posted 2025-09-18 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2023-02

CONDITIONS: Immunomodulatory Drugs; Tuberculosis
Keywords: Nutrition; tuberculosis; immunomodulatory; mushrooms; fortified
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Control group (Placebo Comparator): Patients took Myrin P Fort
  Interventions: Dietary Supplement: Myrin P Fort
- Zn + Se supplemented cookies (Experimental): patients took Zn + Se supplemented cookies
  Interventions: Dietary Supplement: Zn + Se + Myrin P Fort
- Zn + Se + Myrin P Fort (Experimental): Patients took Zn + Se
  + Myrin P Fort
  Interventions: Dietary Supplement: Zn + Se supplemented cookies

INTERVENTIONS:
Dietary Supplement: Myrin P Fort — Patient took Myrin P Fort
  Arms: Control group
Dietary Supplement: Zn + Se supplemented cookies — patients took Zn + Se supplemented cookies
  Arms: Zn + Se + Myrin P Fort
Dietary Supplement: Zn + Se + Myrin P Fort — patients took Zn + Se
  + Myrin P Fort
  Arms: Zn + Se supplemented cookies

SUMMARY:
The primary hypothesis of the study was that zinc and selenium supplementation through fortified cookies would enhance the immune response and improve clinical outcomes in tuberculosis patients. For this purpose, a single-blind randomized control trial was carried out to determine the effect of zinc and selenium on the immunomodulatory parameters of tuberculosis approved by the Ethics Committee of the University of Lahore, Pakistan. In the first phase, the proximate and minerals profile of shiitake mushroom was analyzed, and functional cookies were developed fortified with zinc and selenium. In the second phase, 120 tuberculosis patients were divided into four groups (T0, T1, T2 & T3) to assess the impact of supplementation on anthropometric, microbiological, and hematological parameters. Meanwhile, results were statistically examined through Principal component analysis and a heat map of the attributes under research were generated using R-studio (Version 4.2.2). However, results explained that the therapeutic effect of dosage on anthropometric, microbiological, and hematological measurements showed a significant result (p≤0.05), indicating that zinc and selenium may help to modulate the immunological response, and potentially improving the body's ability to resist tuberculosis.

DETAILED DESCRIPTION:
2. Materials and methods 2.1. Procurement of raw materials Shiitake was procured from the departmental store of Lahore and placed in a sealed bag (Zip bag). All the research work was performed at the University of Lahore's Institute of Food Science and Technology

2.2. Fortification of Zn and Se in the rice flour cookies Cookies were made with rice flour samples supplemented with Zn and Se extracted from shiitake mushroom, at concentrations of 100, 150, and 200 mg/kg of cookie dough, according to the usual process outlined by AACC. Butter, sugar, salt, baking powder, egg, ghee and water were used as common ingredients in all treatments, while Zn, and Se extracted from shiitake powder were used as variable ingredients according to the treatments plan given in ST 1. All ingredients were weighed precisely and mixed homogeneously in laboratory mixer bowl for 10 minutes for each treatment group (T0, T1, T2 and T3). After the homogenous mixing, a resting period of 10 to 15 minutes was applied. The dough was converted into a 5mm thick sheet which was cut into cookies using suitable molds. Baking was accomplished at 170°C for 12 to 15 minutes followed by cooling at room temperature. After cooling, cookies were packed in propylene bags. However, each serving (one cookie) in groups T1, T2, and T3 provided an average of 10 mg:10 µg, 15 mg:15 µg, and 20 mg:20 µg of Zn and Se, respectively, as verified by formulation and batch testing. All batches were processed under standardized conditions to ensure ingredient homogeneity and batch to batch uniformity.

Anthropometric measurements, Microbiological and Hematological Parameters were measured 2.4. Statistical Analysis All resulting data were analyzed statistically to test the significance level (p≤0.05) via the completely randomized design (CRD) by using analytical software statistix (version 8.1).

ELIGIBILITY:
Inclusion Criteria

* Patients aged 30-55 years.
* Confirmed diagnosis of pulmonary tuberculosis (Pul-TB) with positive acid-fast bacilli (AFB) in sputum samples.

Exclusion Criteria

* Patients diagnosed with extra-pulmonary TB.
* Patients who had been on anti-TB therapy for more than 2 months prior to enrollment.

Ages: 30 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-07-25 (Actual); Study Completion 2023-07-25 (Actual)

PRIMARY OUTCOMES:
Anthropometric measurements | 5 months
  Body Mass Index was measured. The formula for Body Mass Index (BMI) is: kg/m^2.
Determination of MAC, MAMC, and TSF | 5 months
  The anthropometric measurements of the patients were assessed, including Mid-Arm Circumference (MAC, cm), Mid-Arm Muscle Circumference (MAMC, cm), and Triceps Skinfold Thickness (TSF, mm). These parameters were measured to evaluate the nutritional and muscle status of the patients

SECONDARY OUTCOMES:
Hematological analysis | 5 months
  Hematological analyses were performed, including hemoglobin concentration (g/dL)

CONTACTS AND LOCATIONS:
Locations (1):
- Sana Noreen, Lahore, Pakistan

IPD SHARING:
Plan to Share IPD: No